CLINICAL TRIAL: NCT03109288
Title: Targeting Residual Activity By Precision, Biomarker-Guided Combination Therapies of Multiple Sclerosis (TRAP-MS)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 170083; 17-I-0083
Record Dates: First submitted 2017-04-11; First posted 2017-04-12 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-11-12

CONDITIONS: Multiple Sclerosis
Keywords: Targeted Therapy; Multiple Sclerosis; Biomarkers; Combination Therapy; Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive | interventions — Pioglitazone; Clemastine; Dantrolene; pirfenidone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination Therapy (Experimental): Any two-drug combination of study interventions
  Interventions: Drug: Pioglitazone; Drug: clemastine fumarate; Drug: Dantrolene; Drug: Pirfenidone
- Monotherapy (Experimental): Any of the study Interventions
  Interventions: Drug: Pioglitazone; Drug: clemastine fumarate; Drug: Dantrolene; Drug: Pirfenidone

INTERVENTIONS:
Drug: Pioglitazone — 15-45 mg po qd
Drug: clemastine fumarate — 8 mg/day (divided into 3 doses of 2, 2, and 4 mg)
Drug: Dantrolene — Up to 200 mg/day (divided into 3 doses of 50mg, 50mg, and 100 mg)
Drug: Pirfenidone — Up to 801 mg po tid. Slow titration over weeks based on tolerability:
  267mg po tid x >= 7d 534 mg po tid x >= 7d 801 mg po tid

SUMMARY:
Background:

In people with multiple sclerosis (MS), brain and cerebrospinal fluid (CSF) biomarkers indicate inflammation or disease. Researchers want to see if 4 drugs given alone or combined affect MS biomarkers. They want to see if a change in biomarker levels can predict which drugs a person with MS might respond to.

Objective:

To see if signs of inflammation in CSF help predict a person s response to different drugs.

Eligibility:

People ages 18 and older who:

* Are in protocol 09-I-0032
* Have progressive MS
* Can stand and walk a few steps
* Take an MS drug

Design:

Participants will be screened in protocol 09-I-0032.

Participants will take 1 of the 4 study drugs. Researchers will call after 1 month to see how they are doing. Some will start a second drug. They may take each drug or combination for up to 18 months.

Participants will have 2 visits a year for up to 6 years. Visits include:

* Medical history
* Physical exam
* Blood and heart tests
* X-rays and scans
* Eye exam and tear collection
* Lumbar puncture: A needle inserted between back bones removes some CSF.
* Lymphocytapheresis: Blood is removed through a needle in one arm and run through a machine. The blood is returned through a needle in the other arm.
* A sensor on the forehead records blood flow and oxygen use.
* Participants may get a device for testing at home.

Participants will stop taking the drugs if they have taken 2 drugs together for 18 months or if they do not do well on the drugs.

Participants will be called 3 months later to see how they are doing....

DETAILED DESCRIPTION:
Objective

Multiple inflammatory and neurodegenerative mechanisms drive progression of disability in fully established multiple sclerosis (MS); therefore, it is unlikely that a single therapeutic agent will be curative. Analogous to cardiovascular diseases, effective treatments for evolved MS will likely require individualized combination therapies that target pathogenic processes active in the particular patient. Ability to reliably measure such pathogenic processes in living patients is a prerequisite for a precision-medicine approach to MS.

Using combinatorial cerebrospinal fluid (CSF) biomarkers, we identified and validated molecular diagnostic tests of MS and its progressive stage, tests that correlate with clinical disability and brain atrophy (i.e., molecular tests of MS progression) and tests that predict future rates of disability progression (i.e., molecular tests of MS severity).

These proteomic tests showed that intra-individually heterogeneous processes, different from those that drive MS susceptibility, underlie continuous accumulation of disability and brain atrophy in patients with progressive MS (PMS), or patients with relapsing-remitting (RRMS) treated with current disease-modifying treatments (DMTs). These processes include compartmentalized inflammation, activation of innate immunity such as myeloid lineage, complement and coagulation cascade, toxic astrocytosis, restructuring of the extracellular matrix in the form of fibrosis, and the re-expression (or lack of it) of developmental pathways related to neurogenesis and remyelination. These alternative, likely pathogenic mechanisms are essentially unaffected by current DMTs, consistent with observations of declining efficacy of FDA-approved DMTs with advancing age of MS patients, so that collectively, they offer no benefit on disability progression after age of approximately 53 years. Consequently, the objectives of this protocol are: 1. To develop clinical trial methodology that allows economical screening of prospective therapeutic agents for their efficacy on biological processes related to MS disease severity using CSF biomarkers; 2. To develop knowledge base of intrathecal effects of current DMTs and novel treatments targeting varied mechanisms of MS progression; and 3. To establish and validate framework for development of effective combination therapies for MS via precision-medicine paradigm.

Study population

Subjects with MS who continue to accumulate clinical disability while untreated (e.g., PMS subjects) or on FDA approved immunomodulatory therapies and can travel to NIH every 6 months and undergo serial lumbar punctures (LP).

Design

The protocol has an adaptable workflow that allows simultaneous assessments of multiple therapeutic agents while maximizing potential therapeutic benefit to the studied subjects and providing knowledge necessary for rational development of future combination therapies for MS. The protocol studies drugs whose mechanism of action (MOA) has the potential to inhibit identified processes underlying MS disease severity. Patients will be assigned to one of the drugs that are not contra-indicated based on existing comorbidities and to which the patient has a therapeutic target (e.g., treatment that inhibits activation of myeloid lineage will be assigned only to patients who have elevated CSF biomarkers of myeloid lineage). Longitudinal measurements of CSF biomarkers will determine if the applied treatment(s) exert the desired pharmacodynamic (PD) effects in the intrathecal compartment. Drugs that do not reproducibly effect CSF biomarkers will be dropped from further study (or will be tested in higher dose, if possible), and replaced by new agents under protocol amendments, while drugs with measurable intrathecal PD activity will be combined to evaluate additive or synergistic effects. Subjects who are treated by drugs that were found to be ineffective will be switched to alternative/new drug and their monotherapy or combination therapy period will be restarted with the goal of each subject finishing 18 months of monotherapy and either continuing monotherapy for an additional 18 months or starting a combination therapy for 18 months with effective drugs only. Safety, tolerability, and pilot clinical/imaging efficacy data will evaluate surrogacy of the biomarkers and collect data for power analysis for future definitive trials. The increased understanding of biomarker biology will be utilized to derive process-specific combinatorial biomarkers and biomarker signatures predictive of clinical efficacy.

Outcome measures

Primary outcome will be the change in Combinatorial Weight-adjusted disability scale (CombiWISE) progression at the end of monotherapy + combination therapy period in comparison to projected baseline disability progression. The acquired longitudinal data will be used for assessment of biomarker surrogacy, for identification and validation of PD markers for development of new therapeutic entities and for power analysis of future/definitive clinical trials.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Enrolled in 09-I-0032 protocol.
* Clinically definite MS.
* Age greater than or equal to 18 years at time of study enrollment.
* Expanded Disability Status Scale (EDSS) 1.0-7.5.
* Documented sustained clinical progression of at least 0.5 CombiWISE points/year (measured by greater than or equal to 4 time-points regression analysis of CombiWISE values spanning at least 1.5 years in total).

  * Because currently only NDS utilizes CombiWISE scale, the progression slopes will be determined from NDS protocols: natural history protocol 09-I-0032 or any of the past NDS clinical trials (protocols 09-I-0197, 10-N-0212, 10-N-0125 and 13-I-0088). Consequently, new patients will be screened to this protocol via 09-I-0032 natural history protocol that contains completely overlapping procedures.
  * It is possible that after other MS centers start using CombiWISE scale, this progression criterion may be derived from outside data, as long as they are adequately documented.
* Subjects of childbearing potential must be willing to use a medically acceptable form of birth control, while being treated on this study.
* Patients who desire to continue their current FDA-approved DMTs based on its perceived (partial) therapeutic benefit will be enrolled with the understanding that the underlying FDA-approved therapy must remain stable during this protocol. If patient desires and/or his/her medical condition requires changing FDA-approved DMT during the duration of this protocol, the drugs administered under this protocol will be withdrawn, to establish new baseline of CSF biomarkers under changed therapy, and, if necessary, to establish new progression rate. New baseline of CSF biomarkers on changed therapy can be established after 6 months of new therapy. Because the efficacy of current DMTs decreases with patient s age so that on average, zero percent efficacy on disability progression occurs after age 53 (Weideman, Tapia-Maltos et al. 2017), only those patients who change to higher potency therapy (i.e., treatment escalation) before age 53 will need to repeat the entire process of establishing baseline progression rate: go back to greater than or equal to 1.5 year baseline period on new DMT to verify that the rate of progression remains greater than or equal to 0.5 CombiWISE points/year. Following therapeutic change that occurs before age 53 will be considered treatment escalation: 1. Initiation of any FDA-approved DMT in previously untreated subject or 2. Change from any low potency (i.e., copaxone, teriflunomide, interferon beta preparations, dimethyl or monomethyl fumarate and fingolimod) to any high potency drugs (i.e., natalizumab, ocrelizumab, rituximab, alemtuzumab, siponimod, cladribine, ofatumumab, ozanimod, ublituximab and mitoxantrone). All other therapy changes (i.e., parallel change from low efficacy to low efficacy or from high efficacy to high efficacy, as well as discontinuation of treatment after age 53) will require new CSF baseline (6 months after such therapy change), but will not require 18 months to calculate new CombiWISE slope. After new CSF baseline, and, if necessary, new CombiWISE progression slopes are established, patient can be matched to the same monotherapy or combination therapy regimen they were on before the immunomodulatory DMT change.
* Willing and able to participate in all aspects of the protocol.
* Able and willing to provide informed consent.

EXCLUSION CRITERIA:

* Clinically significant medical disorders that, in the judgment of the investigators, could expose the patient to undue risk of harm or prevent the patient from safely completing all required elements of the study (such as, but not limited to significant cerebrovascular disease, ischemic cardiomyopathy, clotting disorder, other neurodegenerative disorder, substance abuse or significant psychiatric disorder such as depression with suicidal ideations, unable to perform or tolerate MRI examinations).
* Clinically significant medical disorders, other than MS, that require chronic treatment with immunosuppressive or immunomodulatory agents.
* Pregnancy or breastfeeding.
* Abnormal screening/baseline blood tests exceeding any of the limits defined below:

  * Serum alanine transaminase or aspartate transaminase levels which are greater than three times the upper limit of normal values.
  * Total white blood cell count less than 3,000/mm^3.
  * Platelet count less than 85,000/mm^3.
  * Serum creatinine level greater than 2.0 mg/dl and eGFR (glomerular filtration rate) less than 60.
  * Serological evidence of HIV, HTLV-1 or active hepatitis A, B or C.
  * Positive pregnancy test.

Following drug-specific exclusion criteria will be applied when assigning one of the 4 tested agents (these are not exclusions from the trial)

* Pioglitazone

  * Congestive heart failure.
  * History of bladder carcinoma.
  * Type 1 diabetes.
  * Hypersensitivity to the drug.
  * Taking teriflunomide (Aubagio) because of risk of hypoglycemia on this combination.
* Dantrolene

  * Hypersensitivity to the drug.
  * Hepatic impairment/active hepatic disease (cannot be paired with pirfenidone due to risk of cumulative hepatoxicity).
  * Persistent elevation of LFTs.
  * History of previous drug/medication or alcohol-related liver toxicities.
* Pirfenidone

  * Hypersensitivity to the drug.
  * Hepatic impairment/active hepatic disease (cannot be paired with dantrolene due to risk of cumulative hepatoxicity).
  * Persistent elevation of LFTs.
  * Smoking.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2017-08-11 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Primary outcome will be change in CombiWISE progression rate at the end of monotherapy plus combination therapy period in comparison to projected baseline disability progression. | 1.5 years
  CombiWISE will be calculated from EDSS and SNRS scores derived from NeurEx App, to eliminate noise stemming from ambiguities in translating neurological exam to disability scores.

SECONDARY OUTCOMES:
Change in CombiWISE progression rates between baseline and monotherapy phase, monotherapy and combination therapy phase and between different drugs. | 1 year
Safety and tolerability of individual drugs and their combinations | 1 year
Change in the rate of ventricular atrophy between baseline, monotherapy and combination therapy periods, measured by linear regression slopes of greater than or equal to 3 time-points for each period | 1 year
Correlations between change(s) in CSF biomarkers and clinical efficacy (systems biology approach analyzing drugs/combinations separately and combining all drugs/combinations to a single larger cohort; exploratory analysis) | 1 year
Development of new CSF (combinatorial) biomarkers, new clinical scales, new MRI outcomes will be included in exploratory analyses | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bibiana Bielekova, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Kocot J, Kosa P, Ashida S, Pirjanian NA, Goldbach-Mansky R, Peterson K, Fossati V, Holland SM, Bielekova B. Clemastine fumarate accelerates accumulation of disability in progressive multiple sclerosis by enhancing pyroptosis. J Clin Invest. 2025 May 15;135(10):e183941. doi: 10.1172/JCI183941. eCollection 2025 May 15. PMID 40371642
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2017-I-0083.html
- See also: https://go.usa.gov/xP2YY — https://go.usa.gov/xP2YY